CLINICAL TRIAL: NCT03838900
Title: An Observational Study of Individuals With Type 1 Diabetes Using the Loop System for Automated Insulin Delivery
Brief Title: The Loop Observational Study
Acronym: LOS
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Stanford University (Other); Tidepool Project (Unknown); RileyLink (Unknown)
Responsible Party: Sponsor
Other Study IDs: LOOP
Record Dates: First submitted 2018-11-21; First posted 2019-02-12 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Loop; RileyLink; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Individuals who have not started Loop or who have been on Loop fewer than 7 days at the time of enrollment.
  Interventions: Device: Loop
- Cohort B: Participants who have been using Loop 7 or more days at the time of enrollment.
  Interventions: Device: Loop

INTERVENTIONS:
Device: Loop — The Loop System consists of an insulin pump (certain versions of Medtronic insulin pumps) and a Dexcom or Medtronic CGM. The system includes an iPhone with the Loop app and a RileyLink to communicate between the pump and iPhone. An Apple Watch may optionally be used with the system.

SUMMARY:
An observational study to collect data on the efficacy, safety, usability, and quality of life/psychosocial effects of the Loop DIY automated insulin delivery system.

DETAILED DESCRIPTION:
The study will include both adults and youth in the United States, with a recruitment goal of at least 300-1,250 participants. Data to be collected to address the study objective will include CGM metrics; HbA1c; insulin delivery data; carbohydrate data; activity data from HealthKit; self-reported adverse events (e.g., severe hypoglycemia, diabetic ketoacidosis, hospitalizations); self-reported device issues; and psychosocial and user experience/treatment satisfaction surveys.

Online forms will allow participants to report weekly device issues and serious adverse events including severe hypoglycemia, diabetic ketoacidosis, and hospitalizations. General data updates will be obtained after three, six, and 12 months (and every six months thereafter if study participation continues). A fingerstick blood sample will be collected for HbA1c measurement after three months for cohort A and after six and 12 months for both cohorts. Quality-of-life/psychosocial and treatment satisfaction questionnaires will be completed after six and 12 months; new users also will complete questionnaires after 3 months. Virtual focus groups will be completed within the first three months of starting Loop and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Currently have, or have ordered, the hardware devices necessary to use Loop
* Currently use Loop or have plans to start using Loop for insulin delivery
* Willing and able to provide informed consent (or be a parent or other legally authorized representative) and to provide the data and complete questionnaires that are part of the protocol
* Resident of U.S.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals using or planning to use the Loop system
Sampling Method: Non-Probability Sample
Enrollment: 1212 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Measure of Loop Safety by Self-Report of Diabetic Ketoacidosis (DKA) Events | 6 Months
  Number of DKA events and event outcomes on the Adverse Event and Device Issue - Loop survey. DKA events are defined as the development of ketones with a diagnosis of DKA by a medical provider.
Measure of Loop Safety by Self-Report of Severe Hypoglycemic Events | 6 Months
  Number of severe hypoglycemic events and event outcomes on the Adverse Event and Device Issue - Loop survey. Severe hypoglycemia is defined as low blood sugar that affected the individual's ability to think such that they were unable to treat themselves and needed assistance from someone else. The individual may or may not have lost consciousness.
Measure of Loop Safety by Self-Report of Hospitalization Events | 6 Months
  Number of hospitalizations and event outcomes on the Adverse Event and Device Issue - Loop survey.

SECONDARY OUTCOMES:
Measure of Loop Safety by Self-Report of Diabetic Ketoacidosis (DKA) Events | 12 Months
  Number of DKA events and event outcomes on the Adverse Event and Device Issue - Loop survey. DKA events are defined as the development of ketones with a diagnosis of DKA by a medical provider.
Measure of Loop Safety by Self-Report of Severe Hypoglycemic Events | 12 Months
  Number of severe hypoglycemic events and event outcomes on the Adverse Event and Device Issue - Loop survey. Severe hypoglycemia is defined as low blood sugar that affected the individual's ability to think such that they were unable to treat themselves and needed assistance from someone else. The individual may or may not have lost consciousness.
Measure of Loop Safety by Self-Report of Hospitalization Events | 12 Months
  Number of hospitalizations and event outcomes on the Adverse Event and Device Issue - Loop survey.

OTHER OUTCOMES:
Loop Baseline General Data Collection | Enrollment
  Self-report participant's basic information. No scale provided, variable responses.
Summary statistics for CGM metrics | 6 months and 12 months
  Continuous CGM data from participant's Tidepool account.
Loop Additional Form for Current Loop Users | Enrollment (cohort B), 3 Months (cohort A), 6 Months, and 12 Months
  Self-report of participant's use of Loop and Loop related features. No scale provided, variable responses.
LoopHoles Survey | Enrollment (cohort B), 3 Months (cohort A), 6 Months, and 12 Months
  Self-report of participant's patterns of Loop use. No scale provided, variable responses.
Pittsburgh Sleep Quality Index | Enrollment, 3 Months (cohort A), 6 Months, and 12 Months
  Standardized questionnaire and scoring. Usual sleeping habits for past month. Questions 1 - 9. Overall scores range from 0 to 21, with lower values representing better sleep quality.
Satisfaction of diabetes technology. | Enrollment, 3 Months (cohort A), 6 Months, and 12 Months
  Standardized Diabetes Technology Attitudes - 5 with likert scale questions. Each question is scored on a scale of 1 to 5, with a higher score indicating greater satisfaction with diabetes technology.
Automated Insulin Delivery Satisfaction | Enrollment (Cohort B), Month 3 (Cohort A), Month 6, Month 12
  Change in satisfaction of using Loop. Measured using the standardized INSPIRE (Adult, Parent, and Child) questionnaires. The higher the score the more positive the opinion that automated insulin delivery has had a positive impact on the participant's life.
HbA1c | Enrollment, Month 3 (Cohort A), Month 6, Month 12
  Blood sample.
Device issues related to Loop | Weekly from 7 days after enrollment to 12 months
  Weekly self-report of any device issues that interfered with their ability to use Loop on the Adverse Event and Device Issue - Loop survey. No scale provided.
Hypoglycemia Confidence Scale | Enrollment, Month 3 (Cohort A), Month 6, Month 12
  Standardized questionnaire. Confidence of managing hypoglycemia during daily tasks. Overall scores range from 1 to 4, with higher scores indicating greater confidence in managing hypoglycemia.
Hypoglycemia Fear Survey - Worry Scale | Enrollment, Month 3 (Cohort A), Month 6, Month 12
  Standardized survey. Measures level of worry of low blood sugar, for Adult, Parent, and Child. Items are rated on a 5 point Likert scale from 0 to 4. Total scores and sub-scale scores are sum scores of all relative items. For the adult survey, the score ranges from 0-52. For the children's survey, the score ranges from 0-60. For the parent survey, the score ranges from 0-60. A higher score indicates greater fear of hypoglycemia.
Risk Taking Questions | Enrollment, Month 3 (Cohort A), Month 6, Month 12
  Standardized questionnaire about risk taking behavior. Items are scored on a scale of 1 to 10, with a higher score indicating a greater disposition to take risks.
T1-DDS (Management Distress Items) | Enrollment, Month 3 (Cohort A), Month 6, Month 12
  Standardized questionnaire. Feelings about diabetes management. Overall scores range from 1 to 6, with higher scores indicating higher distress over diabetes management.
Device Discontinuation or Non-start Reasons | Up to 12 months, as needed
  No scale questionnaire allowing varied responses about why participant's stopped using Loop or why they never started.
Loop Follow-Up General Data Collection | Month 3 (Cohort A), Month 6, Month 12
  Self-report of participant's basic information. No scale provided, variable responses.

CONTACTS AND LOCATIONS:
Overall Officials: John Lum, MS, Principal Investigator — Jaeb Center for Health Research
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suttiratana SC, Wong JJ, Lanning MS, Dunlap A, Hanes SJ, Hood KK, Lal RA, Naranjo D. Qualitative Study of User Experiences with Loop, an Open-Source Automated Insulin Delivery System. Diabetes Technol Ther. 2022 Jun;24(6):416-423. doi: 10.1089/dia.2021.0485. Epub 2022 May 12. PMID 35099278
- [Derived] Wong JJ, Suttiratana SC, Lal RA, Lum JW, Lanning MS, Dunlap A, Arbiter B, Hanes SJ, Bailey RJ, Hood KK, Naranjo D. Discontinued Use of the Loop Insulin Dosing System: A Mixed-Methods Investigation. Diabetes Technol Ther. 2022 Apr;24(4):241-248. doi: 10.1089/dia.2021.0362. PMID 34780283